CLINICAL TRIAL: NCT06381284
Title: Expediting Myasthenia Gravis (MG) Diagnostic Evaluation: A Novel, Proof-of-Concept for Undiagnosed, Symptomatic Patients That Uses Social Media Targeting and Self-Assessment
Status: Completed | Type: Observational
Sponsor: ZS Associates (Industry)
Collaborators: UCB Pharma (Industry); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ananda Vishnu Pandurangadu, MD, Senior Consultant, ZS Associates
Other Study IDs: MG-001
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis; Neuromuscular Manifestations; Neuromuscular Diseases
Keywords: Social Media; Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis; Neuromuscular Manifestations; Neuromuscular Diseases | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with undiagnosed neuromuscular symptoms
  Interventions: Behavioral: Social media recruitment; Behavioral: Self-Assessment; Behavioral: Follow-up

INTERVENTIONS:
Behavioral: Social media recruitment — Social media users exposed to a variety of paid social media advertisements as a recruitment tool for study enrollment
Behavioral: Self-Assessment — Eligible participants are asked to complete self-administered physical tests to assess inducible fatigue of specific muscle groups
Behavioral: Follow-up — Patients triaged based on their assessed risk of MG are asked to complete recommended follow-up with a clinician to determine presence of myasthenia gravis

SUMMARY:
This is a fully remote, site-less, prospective, observational study enrolling adults in the United States (excluding U.S. territories) with undiagnosed neuromuscular symptoms. The main study objective is to evaluate the feasibility of a social media recruitment campaign tied to a participant reported symptom survey and self-administered physical assessment tool to influence undiagnosed participants to seek care for suspected Myasthenia Gravis (MG).

DETAILED DESCRIPTION:
Participants with undiagnosed neuromuscular symptoms will be targeted via social media paid advertisements to recruit them to our study landing page (weblink: https://bit.ly/unearthrootcause). Two assessment tools were developed by the study team: the Impact of Daily Living (IDL) Survey and the MG Exercise Assessment. Both tools were designed using supporting literature, accepted guidelines, and a rigorous review via a panel of practicing neurologist key opinion leaders experienced in treating MG patients.

Adult participants who don't have specific diagnosed neurologic conditions will first be screened for eligibility based on the results of the IDL survey which will query participants on the presence or absence of habits/symptoms characteristic of MG. Those who qualify will complete the MG Exercise Assessment in which participants are provided video instructions to perform a series of 10 physical tests to examine if specific muscle groups undergo inducible fatigue. The results of the MG Exercise Assessment are reviewed by a neurologist to determine if participants would benefit further from an in-person neurologist evaluation for MG by a provider. Each participant is provided with a report of the neurologist's evaluation. Participants will be followed for 1 year through bimonthly communications to determine if and when they followed up with a clinician and if they received a confirmed diagnosis of myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

* Reside within the 50 states of the United States at the time of enrollment
* Age 19 or older if reside in Nebraska or Alabama, Age 21 or older if reside in Mississippi, Age 18 years or older if reside in any other state
* Active email account
* Fluency in English (spoken / written), as demonstrated by the ability to read and sign the Informed Consent Form

Exclusion Criteria:

* Live in an overseas territory of the United States
* Inability or unwillingness to provide written informed consent
* Diagnosed myasthenia gravis
* Diagnosed multiple sclerosis
* Have speech impairment, eye/arm/leg weakness due to diagnosed brain cancer, or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants who have undiagnosed neuromuscular symptoms
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Social media recruitment feasibility | Enrollment period (4-6weeks)
  Measure the engagement and feasibility metrics of the social media campaign

SECONDARY OUTCOMES:
MG Exercise Assessment Tool validity | 1 year from time of enrollment
  Estimate preliminary measures of validity for the MG Exercise Assessment Tool

OTHER OUTCOMES:
Time to diagnosis | 1 year from time of enrollment
  Evaluate the time to diagnosis for any participant who has a confirmed diagnosis of MG after the completion of the study compared to that reported in literature

CONTACTS AND LOCATIONS:
Overall Officials: Ananda Vishnu Pandurangadu, MD, Principal Investigator — ZS Associates
Locations (1):
- ZS Associates, Evanston, Illinois, United States

REFERENCES:
- See also: Study landing page — http://bit.ly/unearthrootcause